CLINICAL TRIAL: NCT01775683
Title: A Case-control Study to Determine Whether a Screening Measure of Executive Dysfunction, the Quick EXIT, is Predictive of Chronic Homelessness
Brief Title: Can we Predict Chronic Homelessness?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20120651-01H
Record Dates: First submitted 2012-09-25; First posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Cognitive Impairment
Keywords: homelessness
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A - chronically homeless: Men and women, greater than or equal to age 18 years, English-speaking, who are currently homeless and/or housed in an emergency shelter or housing facility for chronically homeless individuals ≥ 6 months.
- Group B - control/formerly homeless: Men and women, greater than or equal to 18 years, English-speaking who are not homeless ≥4 times in the last 3 years and currently living in stable housing ≥ 6 months and in the last 3 years, has been homeless ≤ 1 month

SUMMARY:
Homeless men and women suffer more illness and sooner death compared to housed people. Among the homeless, there is a group that suffers more illness than others. This group is usually homeless for several months, makes up a smaller proportion of homeless people and uses more resources from emergency shelters than other homeless people. Some have asked if a difference in thinking skills explains how people who are homeless for a long time need more help in getting and keeping housing compared to other homeless persons.

In this study, thinking skills that help a person plan and make decisions will be screened among those who have been homeless for a long time and those who were homeless for a short time. If there is a difference, then screening may change how future homeless people get the help they need.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, greater than or equal to 18 years old, English speaking
* Group A: currently homeless and/or housed in an emergency shelter or housing facility for chronically homeless individuals ≥ 6 months
* Group B: not homeless ≥4 times in the last 3 years and currently living in stable housing ≥ 6 months and in the last 3 years, has been homeless ≤ 1 month

Exclusion Criteria:

At the time of testing, individuals with the following characteristics will be excluded:

1. Altered mental status (determined by Nurse Coordinator through participant response to questions regarding orientation to person, place and season - score of at least 2/3 is considered intact mental status).
2. Present intoxication (determined by Nurse Coordinator through participant evaluation of odour, either alcohol or non-beverage alcohol).
3. Currently violent or aggressive towards testers (determined by Nurse Coordinator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Homeless men and women, greater or equal to 18 years, English-speaking, in Ottawa, ON, Canada
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
The Quick EXIT score | Within 2 weeks of recruitment

SECONDARY OUTCOMES:
The Colour Trails test score | Within 2 weeks of recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Claire Vayalumkal, BASc, MD, Principal Investigator — The Ottawa Hospital Rehabilitation Centre
Locations (1):
- The Ottawa Hospital Rehabilitation Centre, Ottawa, Ontario, Canada